CLINICAL TRIAL: NCT03418363
Title: Effect of the Addition of an Oral Androgen (Dehydroepiandrosterone) on Hepatic Globulins in Users of an Antiandrogenic Combined Oral Contraceptive (Ethinyl Estradiol/Drospirenone)
Brief Title: How DHEA Supplements Affect Coagulation in Women Using Birth Control Pills
Acronym: COC+DHEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OHSU IRB# 17651
Record Dates: First submitted 2017-11-03; First posted 2018-02-01 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Contraceptive Usage; Coagulation
Keywords: Oral contraceptives; Venous thromboembolism; androgenic combined oral contraception
MeSH Terms: conditions — Contraception Behavior; Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHEA Oral Capsule (Active Comparator): Subjects will take 100mg DHEA (dehydroepiandrosterone) daily
  Interventions: Dietary Supplement: DHEA Oral Capsule
- Placebo Oral Capsule (Placebo Comparator)
  Interventions: Other: Placebo Oral Capsule

INTERVENTIONS:
Dietary Supplement: DHEA Oral Capsule — Daily 100mg DHEA supplement
  Arms: DHEA Oral Capsule
Other: Placebo Oral Capsule — Daily oral capsule
  Arms: Placebo Oral Capsule

SUMMARY:
A randomized study is to learn more about how a supplement called DHEA (dehydroepiandrosterone) affects clotting factors in women taking combined oral contraceptive pills. Current research suggests that the progestin hormone in a specific type of birth control pill may increase a woman's blood clot risk. However, it is unknown exactly how the progestin causes the increased risk. This study aims to learn if taking a daily dose of supplemental androgen (dehydroepiandrosterone, or DHEA) in addition to birth control pills containing DRSP affects proteins related to coagulation.

DETAILED DESCRIPTION:
While the pro-thrombotic effects of estrogens are well established in women using combined oral contraception (COC), controversy exists over whether the various synthetic progestogens (progestins) used in combination with ethinyl estradiol in COC formulations may modify the risk of venous thromboembolism (VTE). Several studies have demonstrated that different types of progestins used in COCs influence the magnitude of the estrogen-induced changes in coagulation pathway proteins. However, since hepatocytes do not express progesterone receptor, any activity of a progestin must be indirect. While all progestins on the market are strong agonists for the progesterone receptor (PR), most have variable affinity for the androgen receptor (AR), glucocorticoid receptor (GR), and mineralocorticoid receptor (MR). Generations of progestins have been developed, each successive generation exhibiting decreasing levels of androgenicity. Recent epidemiologic studies have suggested an increased risk of VTE in women using low-androgen progestins relative to those using levonorgestrel-containing products. Although no pattern of hepatic globulin changes has been validated as a surrogate marker for thrombosis risk, the overall magnitude of change in various hepatic proteins involved in coagulation is greater with the newer low-androgenic progestins compared to levonorgestrel, leading some experts to suggest that a progestin's androgenic profile may influence the risk of thrombosis. However, a series of well-designed large prospective cohort studies have not confirmed the increased risk of VTE with low-androgen progestins.

A major problem with reconciling the conflicting results from epidemiologic and prospective studies has been the lack of a clear mechanism, as no studies have demonstrated whether these observed changes are mediated through androgen receptor activity. We hypothesize that androgen receptor activity opposes the estrogen receptor-mediated increase in hepatic clotting factors in women using combined oral contraceptives. To test this hypothesis, we propose a randomized clinical trial in which we will enroll healthy women using combined oral contraception containing ethinyl estradiol (EE) with an antiandrogenic progestin (drospirenone, DRSP). Participants will be randomized to treatment with oral androgen (dehydroepiandrosterone, DHEA) or placebo, and we will collect whole blood samples to measure coagulation pathway-related hepatic globulins (APC-r, Protein S, SHBG) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (18-44 years) in generally good health and with body mass index (BMI) between 18 and 35kg/m2
* Premenopausal, with uterus and at least one ovary intact
* Current users (at least 3 months) of combined oral contraception consisting of 0.02 mg (milligram) ethinyl estradiol and 3 mg drospirenone
* Willing to continue use of current combined oral contraception for the next three menstrual cycles
* Have a prescription for combined oral contraception consisting of ethinyl estradiol and drospirenone for the next four cycles
* Not currently using androgen supplementation
* Willing and able to sign the informed consent
* Willing to comply with the study requirements and visit schedule
* No desire to conceive during study participation, approximately 3 months

Exclusion Criteria:

* Currently enrolled in another clinical trial
* Contraindications to androgen supplementation; history of polycystic ovarian syndrome (PCOS)
* Known or suspected pregnancy, pregnancy within 3 months before study enrollment, or desire to conceive during study participation
* Currently breastfeeding
* Known or suspected alcoholism or drug abuse

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Change in 3-month plasma levels of APC-r | Baseline & Study Completion (month 3)
  Access change in blood levels from baseline (Visit 1) to study completion visit (Visit 2). Collection of whole blood samples from participants to assess change in levels of APC-r after randomization to DHEA supplementation or placebo for 3 cycles (approximately 3 months).
Change in 3-month plasma levels of protein S | Baseline & Study Completion (month 3)
  Access change in blood levels from baseline (Visit 1) to study completion visit (Visit 2). Collection of whole blood samples from participants to assess change in levels of protein S after randomization to DHEA supplementation or placebo for 3 cycles (approximately 3 months).
Change in 3-month serum levels of SHBG | Baseline & Study Completion (month 3)
  Access change in blood levels from baseline (Visit 1) to study completion visit (Visit 2). Collection of whole blood samples from participants to assess change in levels of SHBG after randomization to DHEA supplementation or placebo for 3 cycles (approximately 3 months).
Change in 3-month serum levels of ethinyl estradiol | Baseline & Study Completion (month 3)
  Access change in blood levels from baseline (Visit 1) to study completion visit (Visit 2). Collection of whole blood samples from participants to assess change in levels of ethinyl estradiol after randomization to DHEA supplementation or placebo for 3 cycles (approximately 3 months).
Change in 3-month serum levels of DHEA | Baseline & Study Completion (month 3)
  Access change in blood levels from baseline (Visit 1) to study completion visit (Visit 2). Collection of whole blood samples from participants to assess change in levels of DHEA after randomization to DHEA supplementation or placebo for 3 cycles (approximately 3 months).
Change in 3-month serum levels of free and total testosterone | Baseline & Study Completion (month 3)
  Access change in blood levels from baseline (Visit 1) to study completion visit (Visit 2). Collection of whole blood samples from participants to assess change in levels of total testosterone and free testosterone (calculated using serum albumin) after randomization to DHEA supplementation or placebo for 3 cycles (approximately 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jensen, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States